CLINICAL TRIAL: NCT01367418
Title: Comparison Between Epidural and Patient Controlled Analgesia on Immunological and Inflammatory Systems Following Radical Retropubic Prostatectomy
Brief Title: Effects of Anesthetic Technique on Immune and Inflammatory Systems Following Radical Prostatectomy
Acronym: AIMS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Responsible Party: Principal Investigator, Anil Gupta, Associate Professor, Örebro University, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20110601
Record Dates: First submitted 2011-05-26; First posted 2011-06-07 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Prostate Cancer
Keywords: Analgesia: Thoracic epidural, patient controlled; Surgery: Radical retropubic prostatectomy; Immune system; Inflammation
MeSH Terms: conditions — Prostatic Neoplasms; Inflammation | interventions — Analgesia, Patient-Controlled; Morphine; Tea; Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thoracic Epidural Analgesia (TEA) (Experimental): TEA is used for perioperative pain management, having been used both intra- and postoperatively, up to 48 h.
  Interventions: Drug: Thoracic Epidural Analgesia (TEA)
- Patient controlled analgesia (PCA) (Active Comparator): PCA is the standard of pain management and is usually used for up to 48 h postoperative for pain management following radical prostatectomy.
  Interventions: Drug: Patient controlled analgesia (PCA)

INTERVENTIONS:
Drug: Patient controlled analgesia (PCA) — Morphine 1 mg/ml
  Other Names: Morphine = morphine
  Arms: Patient controlled analgesia (PCA)
Drug: Thoracic Epidural Analgesia (TEA) — Intra-operatively: Bupivacaine 0.5% with adrenaline Post-operatively: Ropivacaine 0.2% + sufentanil 1 ug
  Other Names: Bupivacaine = Marcain; Ropivacaine = Narop; Sufentanil = Sufenta
  Arms: Thoracic Epidural Analgesia (TEA)

SUMMARY:
Several recently published retrospective studies show that regional anaesthesia (RA) can reduce cancer-related mortality following surgical treatment of colorectal, breast and prostate cancers and malignant melanoma. If these results are true, then the choice of perioperative pain management is as beneficial, or even better, than the current oncological therapies. This theory needs to be investigated in a prospective, randomized and controlled trail. We shall perform a prospective, randomized study comparing the effects of Thoracic epidural analgesia (TEA) or patient controlled analgesia (PCA) on postoperative immunological and inflammatory markers in order to understand whether the protective effects, if any, of regional analgesia are due to changes in these markers or whether the underlying mechanisms is not mediated via this stress signalling pathway.

DETAILED DESCRIPTION:
Methods

Thirty patients (ASA status 1-2) in the age group 50 - 75 years, undergoing elective radical retropubic prostatectomy would be included in this pilot study. The exact type of cancer, its staging, degree of spread to proximal or distant sites and the pathologic type of cancer would be recorded. Patients on chronic analgesic medication, endocrinologic and immunologic diseases, those with known allergy to LA and those where epidural catheter placement was contraindicated would be excluded. Patients would be allocated to one of three groups: General anesthesia combined with Epidural anesthesia during and after the operation (Group GE; n = 12), General anesthesia combined with Epidural during anesthesia and local anesthesia postoperatively (Group GL; n = 12), General anesthesia alone (Group GO; n = 10)

Anesthesia and Surgery

All patients would be premedicated with midazolam 0.1 mg/kg 15-30 min before planned surgery, which is a routine in our hospital. Paracetamol 1 g was given orally every 6 h starting with the first dose at the time of premedication. IV access would be attained in the preoperative holding area and further anxiolytic would be given as necessary intravenously.

Epidural technique

In patients in Group GE, an 18 G epidural needle would be inserted at the Th10-12 inter-space using the 'hanging-drop' or loss of resistance technique with the patient in the sitting position in the holding area. The epidural catheter would be inserted and subsequently tested for subarachnoid or intravascular placement using 3 ml of mepivacaine 2% with adrenaline, which is standard practice in our hospital. A bolus dose of 3-4 ml mepivacaine 2% with adrenaline would subsequently be injected and a loss of sensation to cold determined after 10 min. If a sensory block to an upper level of Thoracic 8 dermatome and a minimal lower level of L2 is achieved, the patient would be considered to be ready for induction of anesthesia. If not, a further dose of 2-3 ml mepivacaine 2% with adrenaline would be injected epidurally. If this fails to achieve the desired block, it would be assumed that the catheter was incorrectly placed and the patient offered the choice of one more attempt at epidural catheter placement, or exclusion from the study.

Patients in Group GO would not have an epidural catheter placed. Following transfer to the operating room and routine monitoring, anesthesia would be induced in all patients with fentanyl 2 mg/kg i.v. and propofol 1-2mg/kg until loss of eyelash reflex. Tracheal intubation would be performed after muscle relaxation with rocuronium 0.5 mg/kg and anesthesia maintained with 1-3% sevoflurane and 33% oxygen in air. Mechanical ventilation would be used in a low-flow system in order to maintain an end-tidal CO2 of between 4.5-5.5 kPa. In all patients, sevoflurane concentration would be adjusted in order to maintain adequate anesthetic depth, which would be measured using Auditory evoked potentials (AEP) and maintained between 15-25 (A-line). Tachycardia, despite adequate anesthetic depth, would be treated by giving fentanyl intermittently IV as an analgesic when required during the operation. At the end of surgery, muscle relaxation would be reversed using glycopyrrolate (0.2 mg) and neostigmine (2.5 mg). Radical retropubic prostatectomy would be performed in a standardized way using a lower-abdominal midline incision.

Postoperative Management

During the first 4 h postoperatively, patients in Group GO would receive morphine 1-2 mg IV intermittently for pain relief in the post-anesthesia care unit (PACU) in order that the numeric rating scale (NRS) (0 = no pain, 10 = worst imaginable pain) is < 3. Patients in Group GE would have an infusion of ropivacaine 0.2% 5-10 ml/h epidurally. In the event of pain, morphine (1-2 mg) would be administered intravenously as needed in both groups in order to provide good pain relief and NRS < 3.

All patients would be observed in the PACU for 4 h before being transferred to the general urological ward. The epidural infusion/PCA pump would be continued as long as pain relief is needed using these techniques but for a minimum of 48 h. Subsequently, pain relief would be obtained using oral analgesics using a combination of paracetamol and NSAID drugs.

Recording and Measurements

The total amount of anesthetic and analgesic drugs required during the operation would be recorded. Anesthetic drug requirement would be determined by two methods: end-tidal concentration of sevoflurane recorded every 5 min and the weight of the vaporizer before and after each anesthetic. For all measurements, the time when the anesthetic gases were turned off was considered to be time zero (t = 0). In addition to the routine postoperative protocols, the following measurements were recorded:

Pain intensity: At the site of the incision, 'deep' (visceral) pain and pain on coughing at 1, 4, 12, 24 and 48 h was measured using the NRS.

Rescue analgesic (morphine) consumption: during 0-4 h, 4-24 h and 24-48 h. Supplementary analgesic consumption: Additional analgesics administered in order to relieve pain would be recorded/day.

Side effects: Nausea and/or vomiting (0-4 h, 4-24 h and 24-48 h), pruritus and all other complications were recorded.

Surgical complications: the surgical incision would be inspected daily for evidence of infection and graded as either no evidence of infection (= 0), evidence of inflammation (= 1), mild wound dehiscence or suspected infection (= 2) or pus formation with definite infection (= 3). After 48-72 h, the epidural catheter would be removed and the catheter tip sent for bacterial culture.

Blood sampling:

Patient serum or EDTA/Heparin plasma will be assessed for cytokine levels by a Luminex multiplex assay (Human Inflammation 12-Plex kit; GM.CSF, IFN-g, IL-1b, IL-2, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12, TNF-a and VEGF from R&D system) and PGE2 levels will be measured by an ELISA kit from Cayman Chemicals Company. In addition, markers of systemic inflammatory response, including CRP, white blood cell count, differential count and total platelet count, will also be measured before and after surgery.

Natural Killer (NK) cell activity in the blood would be measured using the FANKIA assay. Clusters of differentiation (CD) markers would be measured.

Stress response would be measured using serum cortisol and prolactin levels.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-2
* Radical retropubic prostatectomy

Exclusion Criteria:

* Chronic use of opiates
* Contraindication to epidural analgesia
* Allergy to component drugs
* Chronic inflammatory diseases
* Use of steroids perioperatively

Ages: 50 Years to 78 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Natural Killer Cell activity | 24 h postoperative
  NK cells are of primary importance in the elimination of tumor target cells at the early stage of tumor development, up to and including tumor metastasis. Decreased NK cell function during the perioperative period is associated with an increased risk of mortality in cancer patients. The NK cell activity would be measured using a special assay called FANKIA

SECONDARY OUTCOMES:
IL-2 | 24 h postoperatively
  Interleucine release is a response to injury and the amount of interleucine in the circulation is related to the degree of trauma. Intensity of trauma is in turn related to the degree of stress response, which is reduced by epidural analgesia
IL-6 | 24 h postoperatively
  Interleucine release is a response to injury and the amount of interleucine in the circulation is related to the degree of trauma. Intensity of trauma is in turn related to the degree of stress response, which is reduced by epidural analgesia
TNF alpha | 24 h postoperatively
  Interleucine release is a response to injury and the amount of interleucine in the circulation is related to the degree of trauma. Intensity of trauma is in turn related to the degree of stress response, which is reduced by epidural analgesia
Serum cortisol | 0 h postoperatively
  Serum cortisol is a marker for stress response which is an important factor in immune response

CONTACTS AND LOCATIONS:
Overall Officials: Anil Gupta, MD PhD, Principal Investigator — Orebro University, Sweden
Locations (1):
- University Hospital, Örebro, Sweden